CLINICAL TRIAL: NCT02080247
Title: A Randomized Controlled Clinical Study Comparing the Efficacy and Safety of Calmoseptine vs Destin Maximum Strength Diaper Rash Paste in Treatment of Incontinence Associated Dermatitis in Older Children and Adults
Brief Title: Treatment of Incontinence Associated Dermatitis in Older Children and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Calmoseptine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPMREB-2012-051-CT-PGH
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Incontinence Associated Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Skin care regimen with Calmoseptine ointment (Active Comparator): In this arm the patients with IAD will receive treatment with Calmoseptine Ointment for 6 days as a part of a structured skin regimen
  Interventions: Drug: Skin care regimen with Calmoseptine ointment
- Control: Skin care regimen with Destin ointment (Active Comparator): In this arm , patient will receive treatment with Destin Maximum Strength 40% Zinc Oxide. Diaper Rash Paste (Destin) for 6 days as part of a structured skin care regimen.
  Interventions: Drug: Skin care regimen with Destin ointment

INTERVENTIONS:
Drug: Skin care regimen with Calmoseptine ointment — Application of Calmoseptine Ointment for 6 days will be applied on the affected area that will be calculated by multiplying the longest portion of the affected area measured in a head to toe orientation by the widest portion of the affected area measured from side to side(in Centimeters).
  Arms: Intervention: Skin care regimen with Calmoseptine ointment
Drug: Skin care regimen with Destin ointment — Application of Destin for 6 days will be applied on the affected area that will be calculated by multiplying the longest portion of the affected area measured in a head to toe orientation by the widest portion of the affected area measured from side to side(in Centimeters). Patients will receive treatment with Destin Maximum Strength 40% Zinc Oxide Diaper Rash Paste (Destin) for 6 days as part of a structured skin care regimen.
  Arms: Control: Skin care regimen with Destin ointment

SUMMARY:
A randomized controlled trial that compared the use of two topical zinc oxide based diaper rash products in a structured care regimen for the treatment of IAD in hospitalized adults and older children.

DETAILED DESCRIPTION:
Patients with IAD were recruited at Philippine General hospital to participate in a randomized controlled trial of two topical zinc oxide based diaper rash products used as part of a structured care regimen. All patients recruited to either arm of the trial received a structured care regimen for treatment of IAD for six days following study entry. At least twice daily and as required by incontinence episodes, treatment and care was provided by nurses and nursing aids trained in the study regimen to ensure its consistent implementation. Wet or soiled diapers were removed and the affected area was gently cleansed. Vigorous cleaning was avoided. A thin layer of the study topical ointment was applied prior to putting on a new diaper. Packs containing all the materials required were prepared for each patient daily, including the same brand of diapers for all patients, skin cleansing products and materials, and the assigned study ointment. Data were collected each day relating to their IAD using the Kennedy Skin Condition Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Participant or next of kin/parent/guardian agree to study inclusion and sign the informed consent form or the assent form according to detailed guidance in the consent / assent section.
* Ages: children (at least 12 years old and up to 18 years old ) and adults (18 years old and above)
* Participant is incontinent* of urine and/or feces and has concomitant Incontinent Associated Dermatitis (IAD). (*Including functional incontinence, whereby the ability to control micturition or defecation is intact, but the patient is unable to toilet normally due to immobilization or other reason.).
* There is a reasonable expectation that the participant will be hospitalized for at least 7 days and will be able to complete the study. (NB Study Participant Withdrawal Criteria b - Any participants discharged from hospital by their attending physician before completion of study participation will automatically be withdrawn from the study. Study participation will not under any circumstances lead to delay in a participant's discharge from hospital.).
* Participant has no known allergy or history of adverse reaction to any of the ingredients in either product or to any topical preparations or skin care products.
* Participant has a diagnosis of IAD with a severity score greater than or equal to 3 as determined by the investigator.

Exclusion Criteria:

* Participant has a pre-existing pressure ulcer of stage 3 or 4 or other full thickness wound within the study area
* Participant has an active dermatological condition, or a history of recurrent dermatological conditions, other than IAD, that may affect healing of IAD or imply difficult healing of IAD. Where uncertainty exists, the Investigators will arrange a consultation with a Consultant Dermatologist
* Participant has any severe acute or chronic medical condition such that trial participation may constitute a risk or may interfere with their medical care or their attending physician advises against participation.
* Participant has in the preceding week been treated with systemic or topical agents (other than topical treatments for IAD) that may affect the IAD healing process (for example steroids).

  e. Participant has a known allergy or previous adverse reactions to any of the ingredients in either product.
* Participant has a diagnosis of IAD with a severity score less than 3 as determined by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Complete healing of Incontinence Associated Dermatitis | 6 days up to complete healing of the Incontinence Associated Dermatitis
  The Primary outcome is complete healing of IAD. Complete healing will be defined with the Kennedy IAD Severity Score. It is a cumulative severity score ranging from zero (no IAD) to 9 (an area > 50 cm² affected, redness or inflammation that is uniformly severe in appearance, extreme erosion of the epidermis and dermis with moderate volume and persistent exudate). The score is generated by the IAD Skin Condition Assessment Tool developed by Kennedy and Lutz, which requires assessors to attribute scores of 0-3 for three domains: size of area affected, skin redness or inflammation, and erosion. The sum of these scores is the IAD Severity Score. The size of IAD affected area will be calculated by multiplying the longest portion of the affected area measured in a head to toe orientation by the widest portion of the affected area measured from side to side (in centimeters). Disposable paper tape measures should be used to prevent cross-infection.

SECONDARY OUTCOMES:
Pain scale measured by Wong Baker | 6 days up to complete healing of the Incontinence Associated Dermatitis
  IAD associated pain will be assessed using Wong Baker pain scale. The Wong Baker scale is the most appropriate pain scale for children or adults with cognitive impairment and VAS for older minors and adults. Wong baker pain scale is a simple visual instrument originally designed for assessing pain in children, but has been used in adult populations.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney B. Dofitas, Medical Doctor, Principal Investigator — University of the Philippines
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, National Capital Region, Philippines

REFERENCES:
- [Derived] Graham T, Beeckman D, Kottner J, Fader M, Fiorentino F, Fitzpatrick JM, Gray M, Harris RG, Sooriah S, Wallace SA, Worsley PR, Woodward S. Skin cleansers and leave-on product interventions for preventing incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2025 Jul 11;7(7):CD011627. doi: 10.1002/14651858.CD011627.pub3. PMID 40643063